CLINICAL TRIAL: NCT03582384
Title: Use of Tocofersolan (Vedrop®) to Prevent or Treat Refractive Vitamin E Deficiency in Infants and Children
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never started
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Daniel Elman, Clinical Research Specialist, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00026926
Record Dates: First submitted 2018-06-26; First posted 2018-07-11 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Short Bowel Syndrome; Vitamin E Deficiency
MeSH Terms: conditions — Short Bowel Syndrome; Vitamin E Deficiency | interventions — tocophersolan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Tocofersolan

INTERVENTIONS:
Drug: Tocofersolan — After baseline labs are obtained, therapy with tocofersolan will be initiated at an initial dose of 17 mg/kg of d-alpha-tocopherol in the form of tocofersolan (0.34 ml/kg/day) and titrated based on blood levels.

SUMMARY:
Patients with short bowel syndrome or other forms of intestinal failure/fat malabsorption are unable to tolerate adequate oral or enteral feedings. They require that nutrition be given as enteral nutrition that is delivered by feeding tube. Often these children take supplements such as vitamins to help improve their nutritional status but, due to their condition, they have difficulty absorbing the supplement sufficiently and most of it is lost in the stool. The drug that will be studied, Tocofersolan (Vedrop®) is a form of vitamin E, a type of the fat soluble vitamin needed in the human diet. It has been formulated in such a way that it may be more easily absorbed by patients with this condition. The main purpose of the study is to learn about the safety and tolerability of this form of vitamin E. Before receiving the study drug, the severity of the child's vitamin E deficiency will be determined by a blood sample, followed by giving them a daily dose of tocofersolan (Vedrop®) either orally or through their feeding tube. After a 4 weeks of therapy, a second blood sample will be checked and the child will continue either same dose of tocoferssolan or it will be adjusted in response to the blood levels. If the study drug works as it is designed to do, there should be an increase in the concentration of the vitamin E in the child's blood, suggesting that the drug was absorbed. At each visit, a sample of blood will be obtained to assess the child's vitamin E status and general health.

Patients will remain on tocofersolan for approximately one year or as long as the study remains open. Based on the European pediatric experience, patients should be expected be on tocofersolan a minimum of 3 months, ideally 6 months to see optimal clinical response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with intestinal failure or fat malabsorption who have refractory vitamin E deficiency (defined as vitamin E level < 5 mg/L) despite receiving vitamin E supplementation with currently available enteral vitamin E products for at least 6 months or requiring the provision of vitamin parenterally as part of a multivitamin infusion.

Exclusion Criteria:

1. Pregnancy
2. Use of warfarin or any related vitamin K antagonist.
3. Enrollment in any other clinical trial involving an investigational agent (unless approved by the principal investigators of the other trial)
4. The parent or guardian or child unwilling to provide consent or assent

Ages: 30 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Vitamin E Level | 1 Year
  Primary outcomes measured will include whether the vitamin E level increased to > 5 mg/L

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Westergren T, Kalikstad B. Dosage and formulation issues: oral vitamin E therapy in children. Eur J Clin Pharmacol. 2010 Feb;66(2):109-18. doi: 10.1007/s00228-009-0729-1. Epub 2009 Oct 13. PMID 19823814
- [Background] European Medicines Agency Evaluation of Medicines for Human Use, CHMP Assessment Report for Vedrop, London, 29 May 2009 Doc.Ref.: EMEA/485798/2009.
- [Background] Sokol RJ. A New Old Treatment for Vitamin E Deficiency in Cholestasis. J Pediatr Gastroenterol Nutr. 2016 Dec;63(6):577-578. doi: 10.1097/MPG.0000000000001330. No abstract available. PMID 27429361
- [Background] Thebaut A, Nemeth A, Le Mouhaer J, Scheenstra R, Baumann U, Koot B, Gottrand F, Houwen R, Monard L, de Micheaux SL, Habes D, Jacquemin E. Oral Tocofersolan Corrects or Prevents Vitamin E Deficiency in Children With Chronic Cholestasis. J Pediatr Gastroenterol Nutr. 2016 Dec;63(6):610-615. doi: 10.1097/MPG.0000000000001331. PMID 27429423
- [Background] Ubesie AC, Kocoshis SA, Mezoff AG, Henderson CJ, Helmrath MA, Cole CR. Multiple micronutrient deficiencies among patients with intestinal failure during and after transition to enteral nutrition. J Pediatr. 2013 Dec;163(6):1692-6. doi: 10.1016/j.jpeds.2013.07.015. Epub 2013 Aug 24. PMID 23978355
- [Background] Zondlo Fiume M. Final report on the safety assessment of Tocopherol, Tocopheryl Acetate, Tocopheryl Linoleate, Tocopheryl Linoleate/Oleate, Tocopheryl Nicotinate, Tocopheryl Succinate, Dioleyl Tocopheryl Methylsilanol, Potassium Ascorbyl Tocopheryl Phosphate, and Tocophersolan. Int J Toxicol. 2002;21 Suppl 3:51-116. doi: 10.1080/10915810290169819. No abstract available. PMID 12537931
- [Background] Ash, M. (2004). Handbook of green chemicals (2nd ed.). Endicott, N.Y.: Synapse Information Resources.
- [Result] Yang CF, Duro D, Zurakowski D, Lee M, Jaksic T, Duggan C. High prevalence of multiple micronutrient deficiencies in children with intestinal failure: a longitudinal study. J Pediatr. 2011 Jul;159(1):39-44.e1. doi: 10.1016/j.jpeds.2010.12.049. Epub 2011 Feb 16. PMID 21324480